CLINICAL TRIAL: NCT03713515
Title: Bridging the Evidence-to-practice Gap: Evaluating Practice Facilitation as a Strategy to Accelerate Translation of a Systems-level Adherence Intervention Into Safety Net Practices
Brief Title: Bridging the Evidence-to-practice Gap
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-01290
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Stepped Wedge
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Faciliation (Experimental): Will be supported by a practice facilitator
  Interventions: Behavioral: ALTA
- Usual Care (No Intervention): Using a stepped wedge design, all practice sites begin as part of the Usual Care (UC) control condition and will receive standard hypertension management that is part of the current clinic procedure. No practice facilitation will occur at this time.

INTERVENTIONS:
Behavioral: ALTA — The study will involve each site starting with the usual care phase, followed by a period of 6 months during which practice facilitators will conduct the pre-implementation evaluation (e.g., workflow analysis, environmental scan), refine the practice facilitation strategies that will be used in the implementation phase, and train staff in the Advancing Medication Adherence for Latinos with Hypertension through a Team-based Care Approach (ALTA) intervention model. ALTA is an efficacious systems-level intervention designed to help patients improve their ability to take their high blood pressure medications and control their blood pressure. Practices and the Project ALTA team will work together to implement the ALTA model into routine care to improve blood pressure control and medication adherence in Latinx patients.
  Arms: Practice Faciliation

SUMMARY:
The proposed project will address this evidence-to-practice gap by evaluating the effect of practice facilitation (PF) of the intervention implementation fidelity (primary outcome) and clinical measures at 12 months (secondary outcomes).

DETAILED DESCRIPTION:
Advancing Medication Adherence for Latinx with Hypertension through a Team-based Care Approach (ALTA) evaluates the effectiveness of using a quality improvement method called practice facilitation (PF) to implement our evidence-based systems-level intervention for improving medication adherence and blood pressure control.

The ALTA intervention focuses on identifying Latinx patients with uncontrolled hypertension who are non-adherent to their antihypertensive medication, referring them to health coaches, coaching patients on medication adherence and self-management, care planning, and monitoring patients to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latino
* Be fluent in English or Spanish
* Be age 18 years or older
* Receiving care in a safety-net primary care practice
* Have uncontrolled HTN documented in the electronic health record (EHR) on at least two visits in the past year (defined as an average BP ≥ 140/90 mmHg)
* Have been prescribed at least one anti-hypertensive medication and be non- adherent to their medications, defined as adherence <80% in the preceding 12 months, as determined by prescription orders obtained from the clinic EHR.

Clinic and nonclinical staff inclusion criteria:

• Primary care provider (MD/DO, NP), Nurse, Medical Assistant, or administrative staff employed at the participating practices and (b) interacts with at least five patients with a diagnosis of hypertension.

Exclusion Criteria:

* Being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks)
* Participation in other hypertension-related clinical trials
* Have significant psychiatric comorbidity or reports of substance abuse (as documented in the EHR)
* Plan to discontinue care at their practice within the next 12 months

Clinic and nonclinical staff exclusion criteria:

• Refuse to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Level of implementation fidelity | 12 months
  Implementation fidelity will be defined as the degree to which ALTA was delivered, as intended. A mixed methods approach will be used to assess the five core domains of implementation fidelity: (1) adherence to the program protocol; (2) dose of the program delivered; (3) quality of program delivery; (4) participant responsiveness; and (5) program differentiation.

SECONDARY OUTCOMES:
Blood Pressure (BP) control | Baseline and 12 months
  First, BP control, will be defined as SBP <140 and DBP <90 mmHg.121 BP control will be assessed using the mean of the last two measurements recorded in the electronic health record (EHR) during each of the pre-intervention and post-intervention study periods (baseline and 12 months). We will also examine the proportion of patients with BP control <130/80 mmHg in exploratory analyses to provide preliminary data on BP control rates of hypertensive Latino patients when considering the new guidelines. We will also explore mean change in systolic and diastolic BP based on the mean of the last two recorded BP readings in the EHR during the pre- and post-intervention periods.
Medication adherence | 12 months
  Will be assessed via pharmacy refills obtained from prescription orders in the clinic EHR using the proportion of days covered (PDC) metric, calculated as the total number of days covered by the medication.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, EdD, Principal Investigator — NYUMC Langone
Locations (1):
- NYUMC Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Access will be granted to Researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided). NYU Data Catalog

REFERENCES:
- [Derived] Chervonski E, Pelegri E, De La Calle F, Mandal S, Graves CA, Colella D, Elmaleh-Sachs A, Nay J, Dapkins I, Schoenthaler A. Cardiovascular Health Markers With Remote Team-Based Hypertension Management in a Safety-Net Population. Am J Prev Med. 2025 Nov;69(5):108031. doi: 10.1016/j.amepre.2025.108031. Epub 2025 Aug 5. PMID 40763829
- [Derived] Schoenthaler A, De La Calle F, De Leon E, Garcia M, Colella D, Nay J, Dapkins I. Application of the FRAME-IS to a multifaceted implementation strategy. BMC Health Serv Res. 2024 Jun 1;24(1):695. doi: 10.1186/s12913-024-11139-0. PMID 38822342
- [Derived] Gago C, De Leon E, Mandal S, de la Calle F, Garcia M, Colella D, Dapkins I, Schoenthaler A. "Hypertension is such a difficult disease to manage": federally qualified health center staff- and leadership-perceived readiness to implement a technology-facilitated team-based hypertension model. Implement Sci Commun. 2024 May 2;5(1):49. doi: 10.1186/s43058-024-00587-8. PMID 38698497
- [Derived] Schoenthaler A, De La Calle F, Leon E, Garcia M, Colella D, Nay J, Dapkins I. Application of the FRAME-IS to a Multifaceted Implementation Strategy. Res Sq [Preprint]. 2024 Feb 12:rs.3.rs-3931349. doi: 10.21203/rs.3.rs-3931349/v1. PMID 38410454
- [Derived] Schoenthaler A, De La Calle F, Soto A, Barrett D, Cruz J, Payano L, Rosado M, Adhikari S, Ogedegbe G, Rosal M. Bridging the evidence-to-practice gap: a stepped-wedge cluster randomized controlled trial evaluating practice facilitation as a strategy to accelerate translation of a multi-level adherence intervention into safety net practices. Implement Sci Commun. 2021 Feb 17;2(1):21. doi: 10.1186/s43058-021-00111-2. PMID 33597041